CLINICAL TRIAL: NCT06850610
Title: Accuracy Of The Owlet OSS 3.0 During Standardized Stable Hypoxia Plateaus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Owlet Baby Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OWL PR0009
Record Dates: First submitted 2025-02-13; First posted 2025-02-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hypoxia
Keywords: hypoxia; pulse oximeter; accuracy; Owlet
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypoxia Plateau Protocol (Experimental): Study participants that all undergo standardized plateaus of oxygen desaturation to evaluate the accuracy of the Owlet noninvasive pulse oximeter during motion and nonmotion conditions.
  Interventions: Diagnostic Test: Pulse oximeter accuracy under hypoxic conditions

INTERVENTIONS:
Diagnostic Test: Pulse oximeter accuracy under hypoxic conditions — This study will specifically evaluate the accuracy of the Owlet pulse oximeter sensor, currently FDA cleared for infants 1-18 months of age in an expanded hypoxia lab trial.

SUMMARY:
This study tests the accuracy of pulse oximeters in a range of arterial oxygen levels from 100% down to 70%. This is done by comparing the test pulse oximeter readings of young, healthy, adult study participants with blood samples drawn from an artery in the wrist during brief plateaus of progressively lower oxygen saturations. The arterial blood sample is processed in a device called a multi-wavelength hemoximeter and compared to the simultaneous oximeter reading. During each set level of oxygen the participant may be asked to have a motion simulator device apply different types of movement to their hands to assess the pulse oximeter's accuracy during motion. This study will be evaluating the Owlet OSS 3.0 sensor, a component in 2 FDA cleared noninvasive pulse oximeters indicated for infants 1-18 months of age.

Testing should require approximately an hour and 15 minutes of the participant's time.

DETAILED DESCRIPTION:
Several separate cohorts of study participants will be recruited and enrolled in accordance with laboratory time and staff availability. After informed consent is performed, a local anesthetic will be injected around the radial artery, and a 22-gauge radial artery catheter will be placed. Pulse oximeters/sensors under test will be attached to the subject along with FDA-cleared reference pulse oximeters. ECG electrodes will be placed on the subject to monitor the subject's heart rate. The Owlet Sensor under test placement and serial numbers will be documented for each subject. Subjects will be placed in a seated, semi-reclined position. Subjects will breathe a nitrogen-air-carbon dioxide mixture to produce the desired level of hypoxemia.

Each subject will undergo two cycles of three different hypoxia plateaus in the 90-100%, 80-90% and 70-80% range, with an average of 20-24 data pairs with a maximum range of 17-30 data points. Study subjects may be have a motion protocol applied to test the Owlet Sensor's accuracy during variable frequencies and amplitudes of movement.

The motions applied by the motion simulator will be 1) 2 Hz sine 10mm 2) 3 Hz sine 10mm 3) 4 Hz sine 10mm 4 ) Random motion 30mm peak, 20 to 200 mm / sec These motions are applied with the fingers tapping on the first cycle of hypoxia and rubbing on the second cycle. The subject will not perform the motion during the first blood sample of each plateau but will during the 2-4th samples separated by 30 seconds.

90% of participants will have at least one usable data point below 85% and at least 69% of subjects will have one usable data pair between 70-80%. As this procedure is evaluating a single user device, a new sensor will be applied to each study participant.

The skin tone distribution of subjects will be divided into 3 groups based on the 10 point Monk skin tone scale (MST) and Individual Typology Angle (ITA) measured by an ISO compliant colorimeter at the forehead and at the anatomic location of sensor placement. MST will be assessed with a printed color swatch that has been verified by a colorimeter. Enrollment of subjects must follow these criteria:

* At least 25% of subjects will be Monk Skin Tone (MST) 1-4 with an ITA greater than 30
* At least 25% of subjects will be MST 5-7 and have an ITA between -30 and 30
* At least 25%-of subjects will be MST 8-10 with an ITA less than -30 (with one half of MST 8-10 subjects having an ITA of less than -50)

ELIGIBILITY:
Inclusion Criteria:

1. The subject is in good general health with no evidence of any medical problems.
2. The subject is fluent in both written and spoken English.
3. The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. The subject is obese (BMI>35).
2. The subject has a known history of heart disease, lung disease, kidney or liver disease.
3. Diagnosis of asthma, sleep apnea, or use of CPAP.
4. The subject has diabetes.
5. The subject has a clotting disorder.
6. The subject has a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
7. The subject has any other serious systemic illness.
8. The subject has a carboxyhemoglobin level greater than 3% (determined during the first sample)
9. Any injury, deformity, or abnormality at the sensor sites that, in the opinion of the investigators' would interfere with the sensors working correctly.
10. The subject has a history of fainting or vasovagal response.
11. The subject has a history of sensitivity to local anesthesia.
12. The subject has a diagnosis of Raynaud's disease.
13. The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
14. The subject is pregnant, lactating or trying to get pregnant.
15. The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
16. The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Pulse Oximeter Accuracy Measures | From enrollment to completion of 6 plateaus of hypoxia over an approximate 75 minute period.
  * Overall Accuracy: Arms is less than 3%.
  * Non-Disparate Performance Evaluation 1: Among pairwise comparisons of MST groups 1-4, 5-7, and 8-10, the largest difference in SpO2 bias is less than 3.5% for the interval 70% ≤ SaO2≤ 85% and less than 1.5% for 85%< SaO2 ≤ 100%.
  * Non-Disparate Performance Evaluation 2: For a 100-point change in emitter sensor site ITA, the difference in SpO2 bias is less than 3.5% for 70% ≤ SaO2≤ 85% and less than 1.5% for 85%< SaO2 ≤ 100%

CONTACTS AND LOCATIONS:
Overall Officials: Koa Gudelunas, Study Director — Vital Signs Research Group
Locations (1):
- Vital Signs Research Group, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data collected during the course of this study are specifically intended for a regulatory submission and may or may not be shared publicly.

REFERENCES:
- [Background] Cohen PR, DiMarco MA, Geller RL, Darrisaw LA. Colorimetric Scale for Skin of Color: A Practical Classification Scale for the Clinical Assessment, Dermatology Management, and Forensic Evaluation of Individuals With Skin of Color. Cureus. 2023 Nov 1;15(11):e48132. doi: 10.7759/cureus.48132. eCollection 2023 Nov. PMID 38046737
- [Background] Bickler PE, Feiner JR, Severinghaus JW. Effects of skin pigmentation on pulse oximeter accuracy at low saturation. Anesthesiology. 2005 Apr;102(4):715-9. doi: 10.1097/00000542-200504000-00004. PMID 15791098
- [Background] Okunlola OE, Lipnick MS, Batchelder PB, Bernstein M, Feiner JR, Bickler PE. Pulse Oximeter Performance, Racial Inequity, and the Work Ahead. Respir Care. 2022 Feb;67(2):252-257. doi: 10.4187/respcare.09795. Epub 2021 Nov 12. PMID 34772785
- [Background] Sjoding MW, Dickson RP, Iwashyna TJ, Gay SE, Valley TS. Racial Bias in Pulse Oximetry Measurement. N Engl J Med. 2020 Dec 17;383(25):2477-2478. doi: 10.1056/NEJMc2029240. No abstract available. PMID 33326721
- See also: A guide to the skin tone stratification used for assessment of accuracy across all represented populations. — https://skintone.google/the-scale